CLINICAL TRIAL: NCT03804866
Title: NGR018: Randomized Phase II Study of NGR-hTNF Plus an Anthracycline Versus an Anthracycline Alone in Platinum-resistant Ovarian Cancer
Brief Title: NGR-hTNF in Combination With an Anthracycline in Platinum-resistant Ovarian Cancer (NGR018)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGR018-IPR/26; 2012-005745-20 (EudraCT Number)
Record Dates: First submitted 2018-10-03; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer
Keywords: NGR-hTNF; Pegylated liposomal doxorubicin; Doxorubicin; Platinum-resistant; Progression or recurrence Ovarian Cancer; Ovarian Cancer; Advanced or metastatic
MeSH Terms: conditions — Ovarian Neoplasms; Disease Progression; Neoplasm Metastasis | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: NGR-hTNF+ anthracycline (Experimental): NGR-hTNF+Pegylated Liposomal Doxorubicin or Doxorubicin
  Interventions: Drug: NGR-hTNF; Drug: Pegylated liposomal doxorubicin; Drug: Doxorubicin
- Arm B: anthracycline (Active Comparator): Pegylated Liposomal Doxorubicin or Doxorubicin
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Doxorubicin

INTERVENTIONS:
Drug: NGR-hTNF — NGR-hTNF: 0.8 mcg/m² as 60 minutes intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs
  Arms: Arm A: NGR-hTNF+ anthracycline
Drug: Pegylated liposomal doxorubicin — 50 mg/m² iv every 4 weeks until confirmed evidence of disease progression
Drug: Doxorubicin — 60 mg/m² iv every 3 weeks for a maximum of 8 cycles

SUMMARY:
The primary objective of this extension protocol is to evaluate the early safety of a new schedule of NGR-hTNF given weekly, instead of every 3 or 4 weeks, in a cohort of 12 patients randomized to the experimental arm A, as compared to a reference cohort of 12 patients randomized to an anthracycline alone

DETAILED DESCRIPTION:
In this extension protocol IPR/26 of completed IPR/24 study, considering the relatively short half-life of approximately 1 hour and the favourable toxicity profile of NGR-hTNF, characterized by transient constitutional symptoms occurring during the first day of administration, an additional cohort of 24 patients will be randomized and the 12 patients enrolled in arm A will receive the same dose of NGR-hTNF 0.8 mcg/m2 given as 60 minutes infusion every week. the weekly schedule of NGR-hTNF 0.8 mcg/m2 has previously been tested in several studies

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically-proven ovarian cancer, fallopian tube and primary peritoneal cancer in advanced or metastatic stage
* Patients previously treated with a maximum of two platinum-based regimen plus paclitaxel and with documented progressive disease on treatment (refractory patient population) or within 6 months from last chemotherapy cycle (resistant patient population)
* ECOG Performance status 0 - 2
* Life expectancy of 12 weeks or more
* Normal cardiac function and absence of uncontrolled hypertension
* Adequate baseline bone marrow, hepatic and renal function defined as follows:

  1. Neutrophils ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL
  2. Bilirubin ≤ 1.5 x ULN
  3. AST and/or ALT ≤ 2.5 x ULN in absence of liver metastasis or ≤ 5 x ULN in presence of liver metastasis
  4. Serum creatinine < 1.5 x ULN
* At least one (not previously irradiated) target lesion or non-measurable disease only, according to RECIST criteria
* Patients may have had prior therapy providing the following conditions are met:

  1. Surgery and radiation therapy: wash-out period of 14 days
  2. Systemic anti-tumor therapy: wash-out period of 21 days
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Patients must not receive any other investigational agents while on study
* More than two previous chemotherapy lines and previous treatment with anthracycline
* Patients with myocardial infarction within the last six months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Prolonged QTc interval (congenital or acquired) > 450 ms
* History or evidence upon physical examination of CNS disease unless adequately treated
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction or contraindications to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety according to NCI-CTCAE criteria (version 4.03) | from the start of treatment until 28 days after last treatment
  To evaluate safety profile related to NGR-hTNF

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | from randomization date, every 6-8 weeks based on chemotherapy during treatment and every 12 weeks during follow-up until first documented PD or death from any cause, whichever came first, assessed up through study completion, approximately 12 months
  Defined as the time from the date of randomization until disease progression, or death
Overall survival (OS) | from randomization date, every 6-8 weeks based on type of chemotherapy during treatment and every 12 weeks during follow-up until date of death, from any cause, assessed up through study completion, approximately 12 months
  defined as the time from the date of randomization until death due to any cause
Response Rate (RR) | from randomization date, every 6-8 weeks based on chemotherapy during treatment and every 12 weeks during follow-up until first documented PD or death from any cause, whichever came first, assessed up through study completion, approximately 12 months
  defined as the percentage of patients who have a best-response rating of complete or partial response, according to standard RECIST criteria
Disease Control Rate (DCR) | from randomization date, every 6-8 weeks based on chemotherapy during treatment and every 12 weeks during follow-up until first documented PD or death from any cause, whichever came first, assessed up through study completion, approximately 12 months
  defined as the percentage of patients who have a best-response rating of complete response, partial response, or stable disease, according to standard RECIST criteria
Duration of Disease Control | from randomization date, every 6-8 weeks based on chemotherapy during treatment and every 12 weeks during follow-up until first documented PD or death from any cause, whichever came first, assessed up through study completion, approximately 12 months
  measured from the date of randomization until disease progression, or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (4):
- Italy (4):
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione "Giovanni Pascale", Naples